CLINICAL TRIAL: NCT06446375
Title: Effects of FIFA 11+ Kids Training Protocol on Motor Competence and Physical Performance in Youth Female Volleyball Players: A Randomized Controlled Trial
Brief Title: FIFA 11+ Kids Training Protocol and Physical Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Nourah Bint Abdulrahman University (Other)
Collaborators: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Monira Aldhahi, Associate professor, Princess Nourah Bint Abdulrahman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023.48.03.07
Record Dates: First submitted 2024-06-01; First posted 2024-06-06 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Athlete; Healthy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental Group (Experimental): FIFA 11+ KIDS Training Protocol will be conducted by the experimental group twice a week for 8 weeks with 15-20-minute interventions. Volleyball players continued their standard volleyball training after the training protocol.
  Interventions: Other: exercise
- Control Group (Active Comparator): The control group will continue their regular volleyball training interventions. All tests were conducted at the same time of day (13:30-16:30) to minimize the impact of circadian rhythms on the results.
  Interventions: Other: Regular daily activity

INTERVENTIONS:
Other: exercise — FIFA 11+ KIDS Training Protocol consists of seven different exercises: three for unilateral, dynamic stability of the lower limbs (hopping, jumping and landing); three for whole body and trunk strength/stability; and one exercise on falling technique.
  Arms: The experimental Group
Other: Regular daily activity — Regular physical activity
  Arms: Control Group

SUMMARY:
This study evaluates the FIFA 11+ Kids Training Protocol, specifically its application to young female volleyball players. It compares it against standard warm-up routines in terms of enhancing motor skills and physical performance. The research anticipates that the FIFA 11+ principles will yield positive outcomes when integrated with existing knowledge of volleyball performance metrics. The study involved 34 young female volleyball players divided into an exercise group (15 players) and a control group (19 players). Initial assessments included anthropometric measurements and motor competence tests such as balancing backward, jumping sideways, moving sideways, and eye-hand coordination (KTK3+ tests).

Subsequent sessions focused on physical and functional tests, including balance performance, agility (pro-agility test), vertical jump (countermovement jump test), and the functional movement screen (FMS) test. A two-way analysis of variance was used to compare the effects of the exercise versus the control group over time, revealing that the exercise group showed significant improvements in dynamic balance, KTK balancing backward, and KTK moving sideways. This study aims to provide innovative insights into the effectiveness of the FIFA 11+ Kids Training Protocol, highlighting its potential benefits in improving physical and motor competencies in young female volleyball players.

DETAILED DESCRIPTION:
Although direct studies on the FIFA 11+ Kids Training Protocol specifically for young female volleyball players are scarce, the program's principles are anticipated to enhance motor skills and physical performance. This study seeks to investigate the potential benefits of applying the FIFA 11+ principles, along with existing insights into motor skills and physical performance in volleyball, to young female players. The objective is to assess how the FIFA 11+ Kids Training Protocol affects motor competence and physical performance. This research aspect is expected to contribute innovative findings to existing literature. The study aimed to determine the effects of the FIFA 11+Kids warm-up program and standard warm-up program on motor competence and physical performance elements of young female volleyball players. A total of 34 volleyball players will complete all the measurement and exercise processes and participate in the post-tests. The experimental design involved participants being randomly assigned to exercise (EG; n=15) and control (CG; n=19) groups. In the first session, anthropometric measurements, including height and body weight, will be measured. Following that, motor competence tests, namely balancing backward, jumping sideways, moving sideways, and eye-hand coordination tests (KTK3+), were measured sequentially. On the second session, physical and functional tests were conducted. These included balance performance measurements, agility test (pro-agility), vertical jump test (countermovement jump test), and functional movement screen (FMS) test. The two-way analysis of variance will be conducted to determine whether being in the exercise group had a significant effect on test scores for mixed measurements, the group-time interaction showed that the exercise group's score increase was significantly higher than that of the control group in dynamic balance, KTK balancing backward and KTK movie sideways parameters

ELIGIBILITY:
Inclusion Criteria:

* Children between age of 11 -13 years old
* typically developing children
* participants should not be using any medication
* Free of any history of cardiovascular disease

Exclusion Criteria:

* Intake of performance-enhancing drugs, anabolic steroids
* Any history of injury, or physiological or physical limitations that could affect the ability to perform training and physical testing in the last year.

Ages: 11 Years to 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Peak power and jump height measurement | at baseline and end of 8 week
  Countermovement Jump (CMJ) values of all participants will be measured. Peak muscle power measures in watts (W) using portable force platform system (peak power2.0, USA). The measurement frequency of the device was set to 500 Hz. Participants will undrergo a 10-minute warm-up program before completing a CMJ. Participants will be asked to begin a downward movement and jump as high as possible after hearing a tone from the computer.
The Body coordination test | at baseline and end of 8 week
  The Body coordination test for children (KTK3+ test battery, supported by a hand-eye coordination task), will be used to assess children's motor competence. KTK3 measures general gross motor coordination . The test include backward balancing (BB), sideways movement (MS), sideways jumping (JS), and hand-eye coordination task (EHC).
Balance tests | at baseline and end of 8 week
  Static and dynamic balance parameters were assessed using a mobile platform that provides an interactive training tool.Participants performed measurements of static and dynamic balance parameters on the mobile platform for 30 seconds in two trials. The highest score from the two trials was used in the statistical analysis.
Pro-agility test | at baseline and end of 8 week
  The test course set with markers placed 5 yards (4.57m) to the left and right of the starting line, with indicators (motivational for the participants' age) placed accordingly. A photocell gate was placed at the starting line to record repeated passage times. Before the start of the application, the participant took their position at the starting line. When ready, they touched the marker on the right first, then the marker on the left, and finally crossed the starting line to finish the test. Measurements will be conducted in two trials.
Functional Movement Screen Test Protocol | at baseline and end of 8 week
  The Functional Movement Screening (FMS)™ system, developed by Gray Cook, Lee Burton and Keith Fields, is a system used to determine potential injury risk in athletes and the quality of individuals' movement patterns, to assess poor neuromuscular control and to improve athletic performance. The Functional Movement Screening test consists of 7 different basic movements (deep squat, hurdle step, single line step, shoulder mobility, active straight leg raise, trunk stability push-up, rotation stability). Scoring for FMS consists of four different possibilities. Scores range from zero to three, with three being the best possible score. The maximum score for the FMS test is 21.

CONTACTS AND LOCATIONS:
Locations (1):
- Monira Aldhahi, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No